CLINICAL TRIAL: NCT07061392
Title: The Effect of Stoma Education Given to Nurses With Two Different Methods on Their Meaningful Learning Self-Awareness, Perceived Learning and Stoma Care Skill Levels: A Randomized Controlled Experimental Study
Brief Title: Stoma Education Methods and Nurse Learning Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve BEKE, Educator Nurse, MsC, PhD, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2024-KAEK-07
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stoma Care Knowledge and Skills of Nurses; Simulation Based Learning; Standardized Patient; Nurse; Self Awareness
Keywords: stoma; nurses; self awarness; meaningful learning; clinical simulation; standardized patients; low reality model

STUDY DESIGN:
Intervention Model Description: The goal of this randomized, parallel-group, assessor-blinded interventional trial was to determine whether stoma-care training using standardized patients, as compared with low-fidelity mannequins, produced superior gains in meaningful learning self-awareness, perceived learning, and practical stoma-care skill levels among oncology nurses at a 600-bed tertiary oncology education and research hospital in Ankara, Turkey.
  Key features of the interventional study model included:
  Design: Two-arm, parallel assignment, assessor-blinded randomized controlled trial.
  Randomization: Ninety nurses were allocated 1:1 to Group M (standardized patient) or Group K (low-fidelity mannequin) using simple block randomization with allocation concealment via sealed envelopes matched to a password-protected Excel list.
  Sample size and flow: Based on G*Power analysis (effect size = 0.6, α = 0.05, β = 0.20), a minimum of 42 nurses per group was required; 45 were enrolled in each arm. After excluding those
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In this trial, the educators who delivered the interventions, the research staff who collected the data, and the investigators who performed the analyses were all aware of participants' group assignments. Only the independent outcome assessor remained blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Group M) (Experimental): Participants in Group M (45 enrolled; 43 analyzed) completed baseline assessments of meaningful learning self-awareness, perceived learning, stoma-care skills, and demographics. They attended a two-hour didactic session on stoma indications, perioperative care, and evidence-based practices. Immediately after, each nurse engaged in a two-hour standardized-patient simulation using realistic stoma moulage. Simulations followed INACSL standards, including a 15-minute pre-briefing, ~20-minute individual in-scenario practice with cueing, peer observation, and a 15-20-minute PEARLS debriefing. All outcome measures were repeated immediately post-training to evaluate short-term cognitive and technical gains.
  Interventions: Other: a low-fidelity Prestan 2000 adult CPR mannequin modified with a play-dough stoma model
- Control Arm (Group K) (Experimental): Group K participants (n = 45 enrolled; 44 analyzed) completed baseline assessments of meaningful learning self-awareness, perceived learning, stoma-care skills, and demographics, and attended the same two-hour didactic session as Group M. They then performed a two-hour stoma-care simulation in small groups on a low-fidelity Prestan 2000 CPR mannequin fitted with a play-dough stoma model. Sessions followed INACSL structure: a brief pre-briefing of objectives and materials; individual mannequin practice with cueing; peer observation in an adjacent area; and a PEARLS-guided debriefing. Outcome measures were repeated immediately post-training to assess short-term cognitive and technical performance.
  Interventions: Other: standardized-patient simulation

INTERVENTIONS:
Other: standardized-patient simulation — Intervention Arm (Group M) Participants randomized to Group M (n = 45 enrolled; 43 analyzed) first completed baseline assessments of meaningful learning self-awareness , perceived learning, and stoma-care skill , as well as a 10-item demographic survey. They then attended a two-hour didactic session-covering stoma indications, types, perioperative care, evidence-based practices, complications, and the stoma-care nurse's role-delivered by a certified stoma-care nurse in small groups.
  Immediately following the lecture, each nurse participated in a two-hour hands-on simulation with a trained standardized patient. The standardized patient had been prepared with a realistic stoma moulage (transparent drape and egg-biscuit mixture) and received two hours of role-training. Simulation sessions adhered to INACSL Standards ("pre-briefing," "in-scenario," "observation," and "debrief
  Arms: Control Arm (Group K)
Other: a low-fidelity Prestan 2000 adult CPR mannequin modified with a play-dough stoma model — Control Arm (Group K) Participants randomized to Group K (n = 45 enrolled; 44 analyzed) underwent the identical sequence of baseline assessments and the same two-hour didactic session as Group M. For the practical component, they performed stoma-care simulation on a low-fidelity Prestan 2000 adult CPR mannequin modified with a play-dough stoma model.
  Hands-on practice was structured in small groups over two hours and included:
  Pre-briefing: Overview of objectives and materials.
  In-scenario: Individual stoma-care performance on the mannequin, guided by the certified stoma-care nurse with cueing as needed.
  Observation: Peers observed from a separate area with scenario summaries.
  Debriefing: Reflection and feedback using the PEARLS framework to consolidate learning and discuss transfer to clinical practice.
  Immediate post-training assessments using the same three scales captured outcomes in meaningful learning self-awareness, perceived learning, and stoma-care skill level.
  Arms: Intervention Arm (Group M)

SUMMARY:
The goal of this randomized controlled trial was to determine whether stoma-care training using standardized patients, as compared with low-fidelity mannequins, improved meaningful learning self-awareness, perceived learning, and practical stoma-care skill levels in oncology nurses at a 600-bed tertiary oncology education and research hospital in Ankara, Turkey. The main questions it aimed to answer were:

Did standardized-patient simulation produce greater gains in meaningful learning self-awareness?

Did it yield higher perceived learning scores?

Did it result in larger improvements in stoma-care skill levels?

Researchers compared Group M (standardized patient) to Group K (low-fidelity mannequin) to evaluate which method more effectively enhanced nurses' cognitive and technical outcomes.

Participants completed a 10-item demographic and background survey, answered pre-training assessments on all three scales, attended a two-hour didactic session on stoma fundamentals and evidence-based care, received two hours of hands-on practice with their assigned modality, and completed immediate post-training assessments using the same instruments.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing graduate
* Working as a nurse in an oncology hospital for at least one year
* Working in inpatient units
* Actively providing care to patients with ostomies

Exclusion Criteria:

* Holding a managerial position
* Having taken a course or received certification on stoma care within the last six months
* Being pregnant, on unpaid leave, or on sick leave
* Participating in another study during the same period
* Incomplete completion of the data collection form
* Voluntary withdrawal from the study during the research period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
practical stoma-care competence | At baseline and immediately after training
  1. Meaningful Learning Self-Awareness Change in total and subscale scores on the 24-item Meaningful Learning Self-Awareness Scale, assessed before and immediately after training. The scale was administered as a self-report questionnaire. Higher post-training scores indicate increased awareness of metacognitive strategies and more effective transfer of learning.
  2. Perceived Learning Change in total and factor scores on the 9-item Perceived Learning Scale, administered before and immediately after training. The scale measures self-perceived learning in cognitive, emotional, and psychomotor domains. Higher post-training scores reflect increased perceived learning gains.
  3. Stoma-Care Skill Proficiency
  Description:
  Change in total scores on the 23-item Stoma Care Skill Rubric, based on direct observation before and immediately after training during simulated stoma-care performance. Higher post-training scores indicate improved technical competence in ostomy care.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Beke, MsC, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided